CLINICAL TRIAL: NCT00509847
Title: A Phase-IIa, Double-blind, Randomized, Controlled Study on the Tolerability and Early Efficacy of hLF1-11 in Hospitalized Patients With Bacteremia Due to Staphylococcus Epidermidis
Brief Title: A Study on the Tolerability and Early Efficacy of hLF1-11 in Patients With Bacteremia Due to S. Epidermidis
Acronym: LIST
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: conduct (recruitment) not feasible within timeframe
Sponsor: AM-Pharma (Industry)
Responsible Party: Dr J Arend, MD, AM-Pharma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMP SSTI 01-01
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2010-01

CONDITIONS: Staphylococcal Infections; Bacteremia
Keywords: S. epidermidis; Staphylococcus; Lactoferrin; hLF1-11; Bacteraemia
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia; Toxemia | interventions — lactoferrin (1-11), human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: human lactoferrin peptide 1-11 — (A) hLF1-11 (once-daily 0.5mg IV for 10 days): Group #1, n=10; OR (B) Placebo (to match hLF1-11): Group #2, n=10
  Other Names: hLF1-11

SUMMARY:
The purpose of this study is to establish the tolerability of treatment with human lactoferrin 1-11 peptide (hLF1-11) administered intravenously as a single dose given for 10 consecutive days, to patients with bacteremia due to staphylococcus epidermidis.

DETAILED DESCRIPTION:
RATIONALE FOR THE STUDY

Choice of Drug

Staphylococcus epidermidis is a relatively uncommon find in blood cultures, most cases being found in patients with intravenous lines through contiguous contamination and current clinical practice is often one of not using antibiotic treatment immediately, unless significant clinical signs and symptoms and/or patient status justifies intervention with an antibiotic. The latter tends to be vancomycin as many S epidermidis strains are resistant to other agents.

hLF1-11 is hypothesized to have antibacterial effects against Staphylococcus epidermidis, amongst other strains.

Should hLF1-11 be shown to be an effective antibacterial against Staphylococcus epidermidis, its use would be justified in other more serious hospital-acquired infections such as MRSA for which hLF1-11 has been shown (in preclinical in vitro and in vivo data) to display a strong therapeutic effect.

Choice of Patient Population

Based on preclinical data hLF1-11 has been shown to possess antibacterial effects on the selected bacteria (Staphylococcus epidermidis). Staphylococcus epidermidis is a commensal found in human skin. In current clinical practice hospital-acquired systemic Staphylococcal epidermidis is not routinely treated unless the bacteremia is accompanied by a clear clinical risk to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with positive blood culture for Staphylococcus epidermidis.
* Diagnosis of staphylococcal infection based on a positive culture for Staphylococcus epidermidis on 2 consecutive occasions within 12 hours.
* Study medication must be started not later than 24 hours of the last qualifying positive blood culture.
* Patients for whom antibiotic treatment is not clinically indicated at the start of the study.
* Patients must have sufficient venous access to permit administration of study drug and monitoring of safety variables.
* Patients who have hepatic and renal parameters within 2X ULN (upper level of normality) at screening.
* Fecund females patients must not be pregnant (confirmed by pregnancy test at entry) and must be on appropriate mechanical (intra-uterine device) or pharmacological ("pill") contraception.
* Written informed consent must be obtained before admission in the study.

Exclusion Criteria:

* Prior antibiotic usage: patients who have received (within 48 hours of study entry) a systemic anti-staphylococcal antibiotic for longer than 24 hours.
* Concomitant antibiotic or anti-bacterial agents except as allowed by the protocol or in life-threatening complications.
* Patients with devices infected with Staphylococcus epidermidis or other important pathogens, including in implants, heart valves and catheters.
* Patients known to have AIDS or who are HIV-positive.
* Neutropenic patients with neutrophil count below 0.5x10^9/L.
* Patients with staphylococcal endocarditis, mediastinitis, meningitis, osteomyelitis and/or joint infections, lung/pleural infections, septic shock.
* Patients with methicillin-sensitive coagulase-negative staphylococcus (CNS) infections (MSSE).
* Patients who have known hypersensitivity to any constituent of hLF1-11.
* Patients who have received an investigational drug within three months prior to the study that may interfere with the interpretation of study results.
* Patients with a concomitant medical condition, in whom, in the opinion of the Investigator, participation may create an unacceptable risk for the patient.
* Patients considered inappropriate by the PI for enrolment in the study, for any reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Haematology, biochemistry, and microbiological evaluation. Adverse event monitoring | 28 Days

SECONDARY OUTCOMES:
Test of Cure (TOC): Microbiological: eradication of Staphylococcus epidermidis bacteria identified at baseline; and Clinical: complete resolution of any clinical signs and symptoms related to bacteraemia due to Staphylococcus epidermidis | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Professor P.E. Verweij, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- UMC St. Radboud, Nijmegen, Gelderland, Netherlands

REFERENCES:
- See also: Related Info — http://www.am-pharma.com